CLINICAL TRIAL: NCT07243353
Title: Examination of the Effect of Nd:YAG Laser on Oxidative Stress and Matrix Metalloproteinase-9 in Teeth With Apical Periodontitis
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ali Turkyilmaz, Associate Professor, Kırıkkale University
Other Study IDs: 2024/046
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Apical Periodontitis; Oxidative Stress
Keywords: Apical periodontitis; Matrix metalloproteinase-9; Nd:YAG laser; Oxidative stress
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nd:YAG laser group: Group treated with Nd:YAG laser
- Control group: Group not treated with Nd:YAG laser

SUMMARY:
The objective of this clinical investigation is to examine the impact of Nd:YAG laser therapy on oxidative stress and matrix metalloproteinase-9 (MMP-9) levels in teeth afflicted with apical periodontitis. Samples were collected from patients who had undergone treatment with the Nd:YAG laser and compared with samples collected from patients who had not received this treatment. The study commenced with a sample of 60 patients. However, the study was completed with 58 patients. The study concluded with the following finding: the use of Nd:YAG lasers was not found to be superior.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 25 and 50 years and classified as American Society of Anesthesiologists (ASA) I. The maxillar and mandibular incisors and premolars with chronic apical periodontitis of a PAI score of 3 or 4 were included.

Exclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) classification II or higher, pregnant, patients with localised or generalised periodontitis, patients who had used antibiotics in the last month and anti-inflammatory drugs in the last week, smokers, and teeth with internal or external root resorption, swelling, palpation pain or fistula in the relevant area, root fracture or incomplete root formation, and teeth that could not be isolated with rubber dam were not included in the study.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — biologically male and female patients
Study Population: The study groups comprised of patients who had applied to the Department of Endodontics at the Faculty of Dentistry at Kırıkkale University and that underwent endodontic treatment from 15 February 2024 to 15 October 2024.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Measurement of TOS, TAOC and MMP-9 levels in periapical exudate and GCF | The initial and seventh days of the treatment period
  TOS, TAOC and MMP-9 levels were measured by ELISA in periapical exudate and GCF samples collected during routine root canal treatment in patients with apical periodontitis. No significant difference was detected in the change in biomarker levels between the group treated with the Nd:YAG laser and the control group.

SECONDARY OUTCOMES:
Determination of the correlation relationship between TOS, TAOC and MMP-9 levels in periapical exudate and GCF samples | The initial and seventh days of the treatment period
  The present study investigated the correlation between periapical exudate and GCF samples. The findings revealed a unidirectional and strong relationship between TOS and TAOC.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale Üniversitesi Diş Hekimliği Fakültesi, Kırıkkale, Turkey (Türkiye)